CLINICAL TRIAL: NCT02068781
Title: Aldosterone-induced Microvascular Dysfunction as a Cause of Salt-sensitivity in Obesity?
Brief Title: Aldosterone, Microvascular Function and Salt-sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Monica Schütten, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 47438/IMP10124
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Abdominal Obesity; Metabolic Syndrome; Sodium-sensitivity; Insulin Resistance; Hypertension
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Insulin Resistance; Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Start with low-sodium diet (Active Comparator): One week of low-sodium diet, followed by a two-week wash-out period and subsequently, another week of high-sodium diet
  Interventions: Dietary Supplement: Low-sodium diet; Dietary Supplement: High-sodium diet
- Start with high-sodium diet (Active Comparator): One week of high-sodium diet, followed by a two-week wash-out period and subsequently, another week of low-sodium diet
  Interventions: Dietary Supplement: Low-sodium diet; Dietary Supplement: High-sodium diet

INTERVENTIONS:
Dietary Supplement: Low-sodium diet — 50 mmol NaCl per 24h
Dietary Supplement: High-sodium diet — 250 mmol NaCl per 24h

SUMMARY:
Currently, the incidence of obesity and obesity-related disorders is reaching epidemic proportions, which entails an increasing burden for health care systems. The association of obesity with other risk factors for type 2 diabetes mellitus and cardiovascular disease, such as insulin resistance and hypertension, is often referred to as the metabolic syndrome. During recent years, salt-sensitivity of blood pressure has emerged as an additional cardiovascular risk factor that is related to obesity and other key components of the metabolic syndrome. The underlying pathophysiological mechanisms of these interrelationships are complex and incompletely elucidated. Microvascular dysfunction has been proposed as a link between insulin resistance and hypertension in obese individuals. In addition, impairment of microvascular function was found to be associated with salt-sensitivity of blood pressure. Increased aldosterone levels, as observed in obese individuals, might be a cause of microvascular dysfunction-induced salt-sensitivity and insulin resistance. Aldosterone not only gives rise to sodium-retention in the distal tubule of the kidney, but was also found to impair endothelial function and thus lower NO-availability, which is characteristic of microvascular dysfunction. In addition, elevated aldosterone levels are associated with both hypertension and insulin resistance, which is illustrated in patients with primary aldosteronism, but also in the general population.

The investigators hypothesize that increased aldosterone levels in obese individuals lead to impairment of microvascular function through reduction of NO-availability. This microvascular dysfunction is suggested to play a central role in the pathogenesis of salt-sensitive hypertension and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

Obese individuals

* Age 18-65 years
* Caucasian
* Waist circumference > 102 cm (men)/> 88 cm (women)

Lean individuals

* Age 18-65 years
* Caucasian
* Waist circumference < 94 cm (men)/< 80 cm (women)

Exclusion Criteria:

Obese/lean individuals

* Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, congestive heart failure, cardiac shunts, cardiac surgery, pulmonary hypertension, cardiac arrhythmias, family history of cardiac arrhythmias or sudden cardiac death)
* Diabetes mellitus/impaired glucose metabolism (fasting glucose values > 5.6 mmol/L
* Stage 3 hypertension (blood pressure > 180/110 mm Hg)
* Unstable or severe pulmonary disease
* Unstable or severe thyroid disorders
* Inflammatory diseases
* Smoking
* Alcohol use > 2 U/day (women)/> 3 U/day (men)
* Use of antihypertensive, lipid-lowering or glucose-lowering medications
* Use of corticosteroids and regular use of NSAIDs
* eGFR< 60 mL/min
* Impairment of hepatic function
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Difference in capillary recruitment between low- and high sodium diets | One week low-sodium diet; wash-out period of two weeks; one week high-sodium diet; order of respective diets is randomized

CONTACTS AND LOCATIONS:
Overall Officials: C.D.A. Stehouwer, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Zhou TL, Schutten MTJ, Kroon AA, Henry RMA, Houben AJHM, van der Kallen CJH, van Greevenbroek MMJ, de Leeuw PW, Stehouwer CDA. Urinary Sodium Excretion and Salt Intake Are Not Associated With Blood Pressure Variability in a White General Population. J Am Heart Assoc. 2023 Jan 3;12(1):e026578. doi: 10.1161/JAHA.122.026578. Epub 2022 Dec 24. PMID 36565181
- [Derived] Schutten MT, Kusters YH, Houben AJ, Niessen HE, Op 't Roodt J, Scheijen JL, van de Waardenburg MP, Schalkwijk CG, de Leeuw PW, Stehouwer CD. Glucocorticoids affect metabolic but not muscle microvascular insulin sensitivity following high versus low salt intake. JCI Insight. 2020 Mar 26;5(6):e127530. doi: 10.1172/jci.insight.127530. PMID 32107343